CLINICAL TRIAL: NCT01051778
Title: Low-molecular-weight Heparin Versus Unfractionated Heparin in Pregnant Women With History of Recurrent Abortion Secondary to Antiphospholipid Syndrome. A Randomized Controlled Trial
Brief Title: Low-molecular-weight Heparin (LMWH) Versus Unfractionated Heparin (UFH) in Pregnant Women With Recurrent Abortion Secondary to Antiphospholipid Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Ahmed Elgazzar Hospital (Other)
Responsible Party: Usama M. Fouda, Ahmed M .Sayed, Cairo university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aps/UFH/enox40
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2010-01

CONDITIONS: Recurrent Abortion
Keywords: Recurrent abortion; Antiphospholipid syndrome; unfractionated heparin; Low Molecular Weight Heparin
MeSH Terms: conditions — Abortion, Habitual; Antiphospholipid Syndrome | interventions — Enoxaparin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enoxaparin 40 mg plus low dose aspirin (Experimental)
  Interventions: Drug: enoxaparin 40mg plus low dose aspirin
- Heparin calcium 5,000 U twice daily plus low dose aspirin (Active Comparator)
  Interventions: Drug: Heparin calcium5,000 U twice daily plus low dose aspirin

INTERVENTIONS:
Drug: enoxaparin 40mg plus low dose aspirin — Enoxaparin 40mg/day by subcutaneous injection ( Clexane 40 mg, Aventis international, Sanofi-aventis France ) is started when the serum pregnancy test become positive. Enoxaparin is stopped 2 days before planned induction of labor or cesarean section and twice-daily unfractionated heparin (UFH) is initiated. The evening UFH dose is cancelled before planned caesarean section . The patients are asked to stop enoxaparin or UFH with the beginning of labor pains . Low dose aspirin (75 mg/day)(Aspocid Paediatric ,Chemical Industries Development (CID)) is started before conception and continued until 36 weeks gestation.
  Other Names: Clexane 40 mg
  Arms: enoxaparin 40 mg plus low dose aspirin
Drug: Heparin calcium5,000 U twice daily plus low dose aspirin — Heparin Calcium 5,000 U twice daily (Cal-Heparine, Amoun Pharmaceutical Co, Egypt) by subcutaneous injection is started when the serum pregnancy test become positive. The evening UFH dose is cancelled before planned caesarean section . The patients are asked to stop UFH with the beginning of labor pains . Low dose aspirin (75 mg/day)(Aspocid Paediatric ,Chemical Industries Development (CID))is started before conception and continued until 36 weeks gestation .
  Other Names: Cal-Heparine
  Arms: Heparin calcium 5,000 U twice daily plus low dose aspirin

SUMMARY:
The aim of this study is to compare the efficacy and safety of Low molecular weight heparin (LMWH) plus low dose aspirin (LDA) with unfractionated heparin(UFH) plus LDA in women with recurrent pregnancy loss associated with antiphospholipid syndrome (APS).

DETAILED DESCRIPTION:
Women with antiphospholipid syndrome (APS) have live birth rates as low as 10% in pregnancies without pharmacological treatment. Low dose aspirin (LDA) ,unfractionated heparin(UFH) , Low molecular weight heparin (LMWH) , prednisone, and intravenous immunoglobulin (IVIG) have been used either alone or in combination in order to improve the live birth rate in APS positive women with recurrent miscarriage. A Cochrane review of 13 randomized or quasi-randomized, controlled trials of various management options of pregnant women with a history of pregnancy loss and APL, revealed that combined UFH and aspirin was the treatment of choice which reduced pregnancy loss by 54% .

During the past decade , low molecular weight heparins were widely used in the prophylaxis and treatment of patients with venous or arterial thrombosis ,with an efficacy and safety superior or at least equivalent to that of UFH .Although recent studies reported the use of LMWH in the management of patients recurrent pregnancy loss secondary to antiphospholipid syndrome resulted in encouraging results . It is not clear whether the efficacy and safety of LMWH is equivalent to that of UFH .

Although LMWH is more expensive than UFH . LMWH has longer half life , greater bioavailability , more stable dose-response relationship than UFH and therefore can be administered once daily. Furthermore, LMWH requires less frequent monitoring than UFH and and has less adverse effect on bone mineral density and platelet count .These advantages make LMWH more attractive for the patients and physicians than UFH .

There are only two studies which compared the efficacy of LMWH plus LDA with that of UFH plus LDA in the management of pregnant women with recurrent pregnancy loss secondary to APS. In addition ,no randomized controlled study has yet compared the efficacy of LMWH plus LDA with UFH plus LDA.

The aim of this study is to compare the efficacy and safety of Low molecular weight heparin (LMWH) plus low dose aspirin (LDA) with unfractionated heparin(UFH) plus LDA in women with recurrent pregnancy loss associated with antiphospholipid syndrome (APS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a minimum of three consecutive pregnancy losses before 10 weeks gestation
* Positive lupus anticoagulant and/or anticardiolipin antibodies (IgG and IgM) on at least two occasions twelve weeks apart .
* Age between 19 - 37 years,
* Body mass index between 19-30

Exclusion Criteria:

* Parental chromosomal abnormalities
* Uterine abnormalities
* Luteal phase defect
* Systemic lupus erythematosus
* Previous thromboembolism
* Sensitivity to aspirin.

Ages: 19 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Principal Investigator — Lecturer of obstetrics and Gynecology , Cairo university; Ahmed M Sayed, Principal Investigator — Assistant professor of obstetrics and Gynecology , Cairo university.
Locations (2):
- Egypt (2):
  - Ahmed Elgazzar hospital, Cairo
  - Cairo university hospital, Cairo

REFERENCES:
- [Background] Noble LS, Kutteh WH, Lashey N, Franklin RD, Herrada J. Antiphospholipid antibodies associated with recurrent pregnancy loss: prospective, multicenter, controlled pilot study comparing treatment with low-molecular-weight heparin versus unfractionated heparin. Fertil Steril. 2005 Mar;83(3):684-90. doi: 10.1016/j.fertnstert.2004.11.002. PMID 15749498
- [Background] Stephenson MD, Ballem PJ, Tsang P, Purkiss S, Ensworth S, Houlihan E, Ensom MH. Treatment of antiphospholipid antibody syndrome (APS) in pregnancy: a randomized pilot trial comparing low molecular weight heparin to unfractionated heparin. J Obstet Gynaecol Can. 2004 Aug;26(8):729-34. doi: 10.1016/s1701-2163(16)30644-2. PMID 15307977
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837
- [Derived] Fouda UM, Sayed AM, Abdou AM, Ramadan DI, Fouda IM, Zaki MM. Enoxaparin versus unfractionated heparin in the management of recurrent abortion secondary to antiphospholipid syndrome. Int J Gynaecol Obstet. 2011 Mar;112(3):211-5. doi: 10.1016/j.ijgo.2010.09.010. Epub 2011 Jan 19. PMID 21251653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between June 2006 to December 2009 at Cairo university hospital and Ahmed Elgazzar hospital ,Cairo.
Period: Overall Study
Arm/Group | Enoxaparin 40 mg /Day Plus Low Dose Aspirin | Heparin Calcium 5,000 U Twice Daily Plus Low Dose Aspirin
Started | 30 (June 2006) | 30 (June 2006)
Completed | 30 (November 2009) | 30 (November 2009)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin 40 mg /Day Plus Low Dose Aspirin | Heparin Calcium 5,000 U Twice Daily Plus Low Dose Aspirin | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.47 (3.20) | 28.57 (3.48) | 28.016 (3.362)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Live Birth Rate = (Number of Live Births / Total Number of Pregnancies)
Description: Live birth occurs when a fetus (> 24 weeks ) , exits the maternal body and subsequently shows signs of life, such as voluntary movement, heartbeat, or pulsation of the umbilical cord.
Time Frame: pregnancy > 24weeks gestation
Measure: Number; unit: Percentage of pregnancies
Arm/Group | Enoxaparin 40 mg /Day Plus Low Dose Aspirin | Heparin Calcium 5,000 U Twice Daily Plus Low Dose Aspirin
Number analyzed (Participants) | 30 | 30
Percentage of pregnancies | 24 | 20

2. Secondary Outcome: Minor and Major Bleeding
Time Frame: Duration of pregnancy and puerperium
Reporting Status: Not Posted

3. Secondary Outcome: Thrombocytopenia
Time Frame: Duration of pregnancy and puerperium
Reporting Status: Not Posted

4. Secondary Outcome: Preeclampsia
Time Frame: Pregnancy > 20 weeks gestation
Reporting Status: Not Posted

5. Secondary Outcome: IUFD
Time Frame: Pregnancy >24 weeks gestation
Reporting Status: Not Posted

6. Secondary Outcome: Preterm Delivery
Time Frame: 24 weeks gestation<Pregnancy <37weeks gestation
Reporting Status: Not Posted

7. Secondary Outcome: Spontaneous Osteoporotic Fractures
Time Frame: Duration of pregnancy and puerperium
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: June 2006 to December 2009
Arm/Group | Enoxaparin 40 mg /Day Plus Low Dose Aspirin | Heparin Calcium 5,000 U Twice Daily Plus Low Dose Aspirin
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin 40 mg /Day Plus Low Dose Aspirin (N=30) | Heparin Calcium 5,000 U Twice Daily Plus Low Dose Aspirin (N=30)
Severe bleeding episodes , e.g antepartum hemorrhage or postpartum hemorrhage (Reproductive system and breast disorders) | 0 (30) | 0 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes